CLINICAL TRIAL: NCT04544462
Title: ANXA5 M2 Haplotyping in IVF Patients and Embryos
Status: Active, not recruiting | Type: Observational
Sponsor: Genomic Prediction Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Genomic Prediction Inc 625
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Infertility; Miscarriage, Recurrent; Pregnancy Complications
MeSH Terms: conditions — Infertility; Abortion, Habitual; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva swabs will be collected from participants. DNA will be extracted and used to screen for the M2 haplotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infertile patients: Patients attending an IVF center for infertility treatment
  Interventions: Other: M2 Test

INTERVENTIONS:
Other: M2 Test — DNA will be extracted from saliva samples obtained from participants. Genetic testing will be performed to screen for the M2 mutation and determine the carrier status of each patient and partner.

SUMMARY:
This study aims to characterize the association between history of pregnancy complications and M2 carrier status in IVF patients and the utility of M2 haplotype preimplantation genetic testing (PGT) in embryos produced by carrier couples. Participants in this study will be screened for the M2 variant. History of pregnancy complications and miscarriages will be studied in order to determine potential associations with M2 carrier-ship.

DETAILED DESCRIPTION:
Patients consenting to participation in the study will receive a saliva collection kit for M2 testing. Genomic Prediction Clinical Laboratory will perform testing and issue a report per routine clinical procedures. Upon completion of issuing a report, the patients' medical records will be obtained from the IVF Center providing care to the patient. Information obtained may include: history of miscarriage, embryo transfer outcomes, preeclampsia, small for gestation age baby, or thrombophilia disorders.

In addition to obtaining records related to history of pregnancy complications, carrier couples will be offered the use of preimplantation genetic testing for M2 carrier status (PGT-M2) in their embryos. Patients electing to perform PGT-M2 will receive PGT-A according to standard clinical practice, along with M2 carrier status.

A total of 500 patients will complete the study and may be recruited from any IVF clinic in the United States. Patients will undergo ovarian hyper-stimulation, oocyte retrieval, fertilization and embryo culture per standard clinical protocol determined by each clinic.

ELIGIBILITY:
Inclusion Criteria:

* All couples above the age of 18

Exclusion Criteria:

* Any case where biological parental DNA is unavailable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All couples above the age of 18 seeking infertility treatment at IVF centers
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
M2 Haplotype frequency | 1 month
  Frequency of carriers of the M2 haplotype attending an IVF center for infertility treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Genomic Prediction Clinical Laboratory, North Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No